CLINICAL TRIAL: NCT05539573
Title: PROVE ACURATE neo2™ - Post Market Safety and Performance Surveillance in Aortic Stenosis
Acronym: PROVE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: National University of Ireland, Galway (Unknown)
Responsible Party: Principal Investigator, Holger Thiele, Prof. Dr., University of Leipzig
Other Study IDs: PROVE
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Aortic Stenosis
Keywords: Transcatheter aortic valve implantation (TAVI); ACURATE neo2™ bioprosthetic aortic valve; ACURATE neo2™ transfemoral delivery system
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Patients with planned transcatheter treatment of severe aortic stenosis with the ACURATE neo2™ aortic bioprosthesis and ACURATE neo2™ transfemoral delivery system.
  Interventions: Device: Planned TAVI with the ACURATE neo2™ aortic bioprosthesis and ACURATE neo2™ transfemoral delivery system.

INTERVENTIONS:
Device: Planned TAVI with the ACURATE neo2™ aortic bioprosthesis and ACURATE neo2™ transfemoral delivery system. — The study will collect data from patients treated with the ACURATE neo2™ and its transfemoral delivery system following standard TAVI practice at each participating center. All patients will be followed to 12 months after the implant procedure. The study is divided into three periods:
  1. Screening period: from screening to enrollment if study criteria are met.
  2. Implantation procedure: immediately pre-implant to 24 hours post-procedure.
  3. Follow-up period: at hospital discharge, at 30 days and at 12 months post-procedure.

SUMMARY:
Aortic valve sclerosis (aortic valve thickening and calcification without pressure gradient) is one of the most common valvular abnormalities in the Western world. Per year, about 1.8-1.9% of these patients develop aortic valve stenosis which will eventually be treated by TAVI (Transcatheter aortic valve implantation).

The purpose of this study is to collect and monitor ongoing safety and performance clinical data of the ACURATE neo2™ aortic bioprosthesis and the ACURATE neo2™ transfemoral delivery system, hereafter referred to as the ACURATE neo2™ and transfemoral delivery system in the context of an observational investigator initiated trial (IIT).

DETAILED DESCRIPTION:
There are four leading causes of valvular aortic valve stenosis, namely: calcific aortic stenosis, congenital aortic valve malformations, rheumatic aortic valve stenosis, and endocarditis. Calcific aortic valve stenosis is a chronic progressive disease, and the predominant cause of aortic valve stenosis in the Western world. Multiple mechanisms influencing the progression of aortic valve stenosis have been identified. However, there is still no sufficient drug therapy to stop or reverse the process.

If high-grade aortic valve stenosis becomes symptomatic, death rates increase up to 50% in 2 years.Many patients with severe and symptomatic aortic stenosis are successfully treated with surgical aortic valve replacement (SAVR), which can reduce symptoms and improve survival. However, up to one-third of symptomatic patients are considered inoperable due to comorbidities and the high risk of surgery. This treatment gap forced the development of less invasive approaches for patients with aortic stenosis considered inoperable and led to the development of TAVI. Later, TAVI has also been considered in the European Society of Cardiology/European Association for Cardio-Thoracic Surgery (ESC/EACTS) 2017 and American Heart Association/American College of Cardiology (AHA/ACC) guidelines for the management of patients with valvular heart disease and intermediate surgical risk and recently, new landmark studies have expanded the use of TAVI into the low surgical risk field.

For the establishment of TAVI as the first line treatment option in lower risk patients, further improvement with regard to adverse outcomes associated with TAVI (e.g. vascular complications, rates of paravalvular leak/aortic regurgitation and the need for permanent pacemakers) will be essential. Therefore, large registries are needed to detect rare events and tendencies in a real-world setting.

The PROVE study will collect baseline, procedural and follow-up data. In addition, it will serve as an imaging library (angiography, echocardiography and cardiac computed tomography) to evaluate the potential advantages and disadvantages of the ACURATE neo2.

ELIGIBILITY:
Inclusion Criteria:

* Planned transcatheter treatment of severe aortic stenosis with the ACURATE neo2™ aortic bioprosthesis and ACURATE neo2™ transfemoral delivery system.
* Age ≥ 18 years of age
* Written informed consent by patient and/or legal representative

Exclusion Criteria:

* Patient is unlikely to be able or willing to follow the investigator's instructions during study participation.
* Patients temporally unable to provide written informed consent (e. g. unconscious emergency patients)
* 3. Patients placed in an institution by official or court order

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from primary care clinics. As the ACURATE neo2™ is approved for use to treat patients with severe aortic stenosis, the inclusion criteria are broad in order to allow the device to be used in an all-comers population and following the instructions for use (IFU).
Sampling Method: Probability Sample
Enrollment: 1043 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause death | through study completion, an average of 1 year
  The individual survival time is calculated from the day of procedure up to death of any cause or up to the last last date on which the patient was known to be alive.

SECONDARY OUTCOMES:
Mortality (count) | through study completion, an average of 1 year
  Numbers by cause and timing period
Mortality (rate) | through study completion, an average of 1 year
  Rates, by cause and timing period
Neurological events (count) | through study completion, an average of 1 year
  Numbers by type, grading and timing
Neurological events (rate) | through study completion, an average of 1 year
  Rates by type, grading and timing
Myocardial infarction (count) | through study completion, an average of 1 year
  Numbers by type
Myocardial infarction (rate) | through study completion, an average of 1 year
  Rates, by type
Re-hospitalization (count) | through study completion, an average of 1 year
  Re-hospitalization yes/no: numbers -> Total number of re-hospitalization per patient, by type
Re-hospitalization (cumulative incidence) | through study completion, an average of 1 year
  Re-hospitalization yes/no: rates Cumulative incidence of first re-hospitalization, by type
Bleeding events (count) | through study completion, an average of 1 year
  Numbers by type
Bleeding events (rate) | through study completion, an average of 1 year
  Rates by type
Transfusions | through study completion, an average of 1 year
  Total number per patient, by timing period
Vascular and access-related complications (count) | through study completion, an average of 1 year
  Numbers by type and severity
Vascular and access-related complications (rate) | through study completion, an average of 1 year
  Rates by type and severity
Cardiac structural complications (count) | through study completion, an average of 1 year
  Numbers by severity
Cardiac structural complications (rate) | through study completion, an average of 1 year
  Rates by severity
Other acute procedural and technical valve related complications (count) | through study completion, an average of 1 year
  Numbers by category and type of clinical presentation
Other acute procedural and technical valve related complications (rate) | through study completion, an average of 1 year
  Rates by category and type of clinical presentation
Conduction disturbances and arrhythmia (count) | through study completion, an average of 1 year
  Numbers by type, timing and duration
Conduction disturbances and arrhythmia (rate) | through study completion, an average of 1 year
  Rates by type, timing and duration
Acute kidney injury (count) | through study completion, an average of 1 year
  Numbers by stage
Acute kidney injury (rate) | through study completion, an average of 1 year
  Rates by stage
Bioprosthetic valve dysfunction (count) | through study completion, an average of 1 year
  Numbers by type
Bioprosthetic valve dysfunction (rate) | through study completion, an average of 1 year
  Rates by type
Clinically significant valve thrombosis (count) | through study completion, an average of 1 year
  Numbers by timing period
Clinically significant valve thrombosis (rate) | through study completion, an average of 1 year
  Rates by timing period
Patient-reported outcomes and health status | through study completion, an average of 1 year
  Kansas City Cardiomyopathy Questionnaire (KCCQ)

OTHER OUTCOMES:
Composite endpoint: technical success | at exit from procedure room
  According to Valve Academic Research Consortium (VARC)-3 criteria
Composite endpoint: device success | at 30 days post procedure
  According to VARC-3 criteria
Early safety | at 30 days post procedure
  Determined at 30 days post procedure
Clinical efficacy | at 12 months post procedure
  Determined at 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Prof. Dr., Principal Investigator — Leipzig University
Locations (27):
- France (2):
  - Jacques Cartier Private Hospital Massy, Massy
  - Centre Cardiologique du Nord Saint-Denis, Saint-Denis
- Germany (21):
  - Universitätsklinikum Augsburg, Augsburg
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Rhön Klinikum, Campus Bad Neustadt, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Schüchtermann-Schiller'sche Kliniken Bad Rothenfelde GmbH & Co. KG, Bad Rothenfelde
  - Deutsches Herzzentrum der Charité, Berlin
  - Universitätsklinikum Köln, Cologne
  - St. Johannes Hospital, Dortmund
  - Herzzentrum Dresden GmbH Universitätsklinik an der TU Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Elisabeth-Krankenhaus, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg - Bad Krozingen, Freiburg im Breisgau
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
  - Heart Center Leipzig at Leipzig University, Leipzig
  - Augustinum, München
  - Deutsches Herzzentrum, München
  - LMU Klinikum der Universität München, München
  - Uniklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
- Lund University, Lund, Sweden
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No